CLINICAL TRIAL: NCT06568198
Title: Modulation Effect of Transcranial Alternating Current Stimulation (tACS) on Chronic Low Back Pain
Brief Title: Modulation Effect of tACS on Chronic Low Back Pain
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Principal Investigator, Jian Kong, Principal investigator, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 2024p001377; 5R01NS129059-02 (NIH)
Record Dates: First submitted 2024-07-29; First posted 2024-08-23 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Chronic Low-back Pain

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- real tACS (Experimental)
  Interventions: Device: Real tACS
- Sham tACS (Sham Comparator)
  Interventions: Device: Sham tACS

INTERVENTIONS:
Device: Real tACS — α-tACS at a frequency of alpha band at S1
  Arms: real tACS
Device: Sham tACS — Sham tACS with no stimulation applied
  Arms: Sham tACS

SUMMARY:
Investigating the modulation effect of tACS

DETAILED DESCRIPTION:
Investigating the modulation effect of one-month Transcranial alternating current stimulation (tACS) for low back pain

ELIGIBILITY:
Inclusion Criteria:

1. Volunteers 18-60 years of age
2. Meet the Classification Criteria of the chronic LBP (having low back pain for more than 6 months)
3. At least 4/10 clinical pain on the 0-10 LBP NRS
4. At least a 10th grade English-reading level; English can be a second language provided that the patients understand all questions used in the assessment measures
5. Meeting the MRI / MEG / EEG screening criteria

Exclusion Criteria:

1. Specific causes of back pain (eg, cancer, fractures, spinal stenosis, infections)
2. Complicated back problems (eg, prior back surgery, medicolegal issues)
3. The intent to undergo surgery during the time of involvement in the study
4. History of cardiac, respiratory, or nervous system disease that, in the investigator's judgment, precludes participation in the study because of a heightened potential for adverse outcome (for example: asthma or claustrophobia)
5. Presence of any contraindications to MRI scanning (for example: cardiac pacemaker, metal implants, claustrophobia, pregnancy, cannot lie still in fMRI scanner)
6. Concomitant autoimmune, chronic, inflammatory, neoplastic, and psychiatric diseases
7. Pregnant or lactating
8. Conditions making study participation difficult (e.g., paralysis, psychoses, or other severe psychological problems as per the judgment of a study investigator during Session 1)
9. Active substance abuse disorders (based on subject self-report and drug test)
10. Regular use of pain medication such as opioids, nonopioid analgesics, coanalgesics, corticosteroids, or immunomodulatory agents
11. Any medical conditions, such as peripheral neuropathy, that could affect the results of QST
12. Current use of psychotropic medication

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-08-25 (Actual); Primary Completion 2028-02-01 (Estimated); Study Completion 2028-02-28 (Estimated)

PRIMARY OUTCOMES:
Alpha activity at rest | Baseline and week 4
  EEG/MEG data will be collected to measure alpha activity.
TC resting state functional connectivity | Baseline and week 4
  fMRI data will be collected to measure resting state functional connectivity.
Numeric Rating Scale (NRS) for pain intensity | Baseline and week 4
  The NRS is a uni-dimensional measure of pain intensity that uses an 11-point numeric scale. We will use it to measure the average low back pain intensity in the past week.

SECONDARY OUTCOMES:
Alpha activity during tonic pressure pain | Baseline and week 4
  EEG/MEG data will be collected during administration of tonic pressure pain to measure alpha activity changes before and after tACS.
TC functional connectivity during tonic pain | Baseline and week 4
  fMRI data will be collected during administration of tonic pressure pain to measure functional connectivity changes before and after tACS.

CONTACTS AND LOCATIONS:
Locations (1):
- Massachusetts General Hospital, Charlestown, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No